CLINICAL TRIAL: NCT05039008
Title: Effectiveness of Physiotherapy Intervention by Restricting Blood Flow in Improving Muscle Strength in Patients With Hemophilic Arthropathy. Randomized Multicenter Clinical Study.
Brief Title: Restricting Blood Flow in Improving Muscle Strength in Patients With Hemophilic Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: He-Blood
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia
Keywords: Hemophilic arthropathy; Blood flow restriction; Physiotherapy; Muscular strength; Muscle activation; Chronic pain; Functionality; Quality of life
MeSH Terms: conditions — Hemophilia A; Chronic Pain | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction group (Experimental): The intervention will last 4 weeks, with a periodicity of 3 weekly sessions (34). In total there will be 12 sessions lasting between 15 and 30 minutes.
  The exercises will be: squats, knee extension and heel elevation (performing 4 sets of 15 repetitions with 30 seconds of rest between sets).
  Interventions: Other: Blood flow restriction
- Control group (No Intervention): The patients included in the control group will not receive any Physiotherapy intervention and will continue with their usual routine, being evaluated in the same periods as the rest of the patients.

INTERVENTIONS:
Other: Blood flow restriction — The intervention protocol will be carried out under the same environmental conditions and, as far as possible, at the same time. The intervention will last 4 weeks, with a periodicity of 3 weekly sessions. In total there will be 12 sessions that will last between 15 and 30 minutes depending on the number of joints affected.
  Arms: Blood flow restriction group

SUMMARY:
Background. The main physical sequela of patients with hemophilia is the development of a progressive, degenerative intra-articular lesion, known as hemophilic arthropathy). This sequela is manifested by chronic pain, limited range of motion, axial abnormalities, and periarticular muscle atrophy.

Objective. To assess the safety and effectiveness of an intervention through blood flow restriction, regarding the frequency of bleeding and the improvement in the perception of muscle activation and strength, functionality, joint pain, joint status and the perception of quality of life in patients with hemophilic arthropathy. knee and ankle.

Study design. Randomized, multicenter, single-blind clinical study. Method. 20patients with hemophilia A and B will be recruited in this study. Patients will be recruited in 3 regions of Spain. The dependent variables will be: bleeding frequency (self-registration), pain (measured with the visual analog scale), joint status (Hemophilia Joint Health Score scale), strength (dynamometer) and range of motion (goniometer). Three evaluations will be carried out: pre-treatment, post-treatment and after a follow-up period of 4 weeks.

Expected results. Observe the safety of blood flow restriction in hemophilia patients. To analyze the efficacy of blood flow restriction in improving muscle strength, joint pain, range of motion, and joint damage in patients with hemophilic knee and ankle arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* Patients with a medical diagnosis of hemophilic ankle and knee arthropathy
* People over 18 years of age
* Patients on prophylactic or on-demand treatment regimen with FVIII / FIX concentrates

Exclusion Criteria:

* Patients with neurological or cognitive disorders that impede understanding of the test.
* Pain free patients
* Amputees, epileptics or patients with severe vision problems
* Patients who are receiving Physiotherapy treatment at the time of the study
* Patients who have not signed the informed consent document

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline hemarthrosis after treatment and at four weeks. | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  A self-registration will be used to evaluate the frequency of bleeding, and thus the safety of the technique. This self-registration will be given to each patient at the beginning of the study and they must fill in the number of hemarthrosis and their main characteristics: date, origin (traumatic or spontaneous) and location (knee or ankle). The self-registration will be delivered to the evaluator in each of the study evaluations (post-treatment and follow-up).

SECONDARY OUTCOMES:
Change from baseline joint pain after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  The visual analog scale will be used to assess the perception of joint pain, being valued with a range of 0 to 10 points (from no pain to the maximum pain suffered or imaginable) in the joints evaluated
Change from baseline muscle strength after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  With a pressure dynamometer (microFET®2 Digital Handheld model) we will measure the strength of the quadriceps and triceps surae. This device measures in Newton the force that the patient exerts in the requested muscular action. The higher the value, the greater the muscle strength. We will carry out the measurements bilaterally. The patient will be asked 4 maximum isometric contractions of 5 seconds, with a rest of 30 seconds between them, against the dynamometer located in the hand of the evaluator
Change from baseline joint status after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Change from knee and ankle joint status during treatment and follow-up period at four weeks. Measurement instrument: Haemophilia Joint Health Score (scale 0-20).
Change from baseline range of motion after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Change from range of movement of knee and ankle during treatment and follow-up period at four weeks. The range of motion of the knee and ankle joint will be measured using a universal goniometer, using the protocol for measuring joint motion described by the American Academy of Orthopaedic Surgeons.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Rubén Cuesta-Barriuso, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No